CLINICAL TRIAL: NCT06810050
Title: Safety and Effectiveness of CGB-500 Topical Ointment with 0.5% and 1% Tofacitinib for the Treatment of Atopic Dermatitis: a Randomized, Dose-Ranging, Vehicle-Controlled, Double-Blind Trial
Brief Title: Phase 2b Safety and Efficacy Study of CGB-500 Topical Ointment with 0.5% and 1% Tofacitnib for Treatment of Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CAGE Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CGB-500-04
Record Dates: First submitted 2025-01-23; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Atopic Dermatitis (AD)
Keywords: Phase 2b study, study the safety and effectiveness of CGB-500 topical ointment with 0.5% and 1% tofacitinib,
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- CGB 500 ointment with 0.5% tofacitinib (Experimental)
  Interventions: Drug: CGB-500 with 0.5% tofacitinib
- CGB 500 ointment with 1% tofacitinib (Experimental)
  Interventions: Drug: CGB-500 Ointment with 1% tofacitinib
- vehicle ointment (Placebo Comparator)
  Interventions: Drug: Vehicle (placebo)

INTERVENTIONS:
Drug: CGB-500 with 0.5% tofacitinib — CGB-500 is a proprietary ointment formulation
  Arms: CGB 500 ointment with 0.5% tofacitinib
Drug: CGB-500 Ointment with 1% tofacitinib — CGB-500 is a proprietary ointment formulation
  Arms: CGB 500 ointment with 1% tofacitinib
Drug: Vehicle (placebo) — placebo ointment
  Arms: vehicle ointment

SUMMARY:
The goal of this clinical trial is to learn if CGB-500 works to treat atopic dermatitis in participants ages 12 and older. The goal is also to learn about the safety of CGB-500. The main questions it aims to answer are:

Does CGB-500 improve atopic dermatitis by decreasing the area affected and the severity of the lesions? What medical problems do participants have when taking CGB500? Researchers will compare CGB-500 to a placebo (a look-alike substance that contains no drug) to see if CGB-500 works to treat atopic dermatitis.

Participants will:

Take CGB-500 or a placebo every day for 8 weeks. Visit the clinic once every 2 weeks for the first month and at the end of 8 weeks.

Keep a diary of when they use the product and complete a form about their symptoms including itching.

DETAILED DESCRIPTION:
The primary objectives of this study:

* To evaluate the safety and tolerability of CGB-500 topical ointment with 0.5% and 1% tofacitinib for the treatment of atopic dermatitis (AD)
* To evaluate the effectiveness of CGB-500 topical ointment with 0.5% and 1% tofacitinib for the treatment of AD

Key trial design:

Intervention Model: Parallel-group Population Type: Pediatric and adult participants Control: Vehicle (without tofacitinib) Population Diagnosis or Condition: Atopic dermatitis Active Comparator: N/A Population Age: ≥ 12 years Trial Intervention Assignment Method: Randomization Site Distribution: US multicenter Number of Arms: 3 Blinding: participants and investigational staff (sponsor, investigator, and evaluators) Number of Participants: 160 to 180

Arms and Duration:

Total duration of trial intervention for each participant: 8 weeks Total duration of trial participation for each participant: Approximately 10 weeks, 2 weeks of screening and 8 weeks of treatment

Arms and Duration Description:

All participants will undergo approximately 2 weeks (Day -15 to Day -1) of screening and 8 weeks of treatment and will be randomized in a 1:1:1 ratio to the following treatment arms. The goal is to randomize 60 participants with a minimum of 48 participants in each of the arms.

* CGB-500 Topical Ointment with 0.5% Tofacitinib BID
* CGB-500 Topical Ointment with 1% Tofacitinib BID
* Vehicle for CGB-500 Topical Ointment BID

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this trial, an individual must meet all of the following criteria:

1. Outpatient, male or female of any race, 12 years of age or older. Females of childbearing potential (FOBCP) must have a negative urine pregnancy test at Screening and Baseline and practice a reliable method of contraception throughout the trial.
2. Have a clinical diagnosis of atopic dermatitis (AD) for at least 12 months prior to Baseline that has been clinically stable disease for ≥ 3 months at the time of the screening visit and prior to dose administration and is confirmed to be AD according to the criteria of Hanifin and Rajka.
3. Have an IGA (Investigator's Global Assessment) score of 2, 3, or 4 at Screening and Baseline.
4. Have AD lesions/symptoms covering at least 1% but less than 10% of total BSA (excluding scalp, genitalia, palms, and soles) at Screening and Baseline.
5. Have at least 1 "target lesion" that measures approximately 10 cm2 or more at Screening and Baseline. Lesion must be representative of the participant's disease state and not be located on the scalp, genitalia, palms, or soles.
6. In general, good health as determined by medical history and physical examination at the time of screening (investigator discretion).
7. Have peak pruritus numeric rating scale (PPNRS) score of ≥ 4 on the scale 0 to 10 at Screening and Baseline.
8. Be able to follow trial instructions and likely to complete all required visits.
9. Sign the institutional review board (IRB)-approved informed consent form (ICF, which includes HIPAA) and assent prior to any trial-related procedures being performed.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this trial:

1. Females who are pregnant, breastfeeding, intending to be pregnant during the trial, or who do not agree to use an acceptable form of birth control during the trial if of childbearing potential .
2. Immunocompromised individuals as adjudicated by the principal investigator (PI) based on review of medical history.
3. Known hypersensitivity or previous allergic reaction to any constituent of the IP (e.g., tofacitinib or Janus kinase (JAK) inhibitors, essential oils, choline, phosphatidylcholine, glycerol, propylene glycol, polyethylene glycol).
4. Has clinically significant safety labs (hematology, chemistry, and urinalysis) at the Screening visit that, in the opinion of the investigator, would preclude participation in the study or affect proper assessment of the study endpoints
5. Skin infections (e.g., bacterial, fungal or viral) that can interfere with reliable AD assessments.
6. Basal cell carcinoma within 6 months prior to Baseline.
7. History of confounding skin conditions, e.g., psoriasis, rosacea, erythroderma, or ichthyosis or presence of Netherton's Syndrome, immunological deficiencies or diseases, HIV, uncontrolled diabetes, malignancy, or serious active or recurrent infection.
8. Known hepatic impairment or disorder and/or ALT and AST >3X ULN at Screening.
9. Has unstable and impaired renal function with an estimated glomerular filtration rate (eGFR) <60 mL/min using Cockcroft-Gault (C-G) equation (eGFR between 60 to <90 mL/minute or higher is acceptable).
10. Use of moderate to strong CYP3A4 and CYP3A5 inhibitors (e.g. ritonavir, clarithromycin, itraconazole, erythromycin, fluconazole, verapamil, ketoconazole, nefazodone, nelfinavir, diltiazem, ciprofloxacin, grapefruit juice) within 4 weeks prior to Baseline.
11. Participants who have previously failed or had an inadequate response to oral, systemic or topical JAK inhibitors, including in a trial or under a prescription for atopic dermatitis (e.g., ruxolitinib, tofacitinib, baricitinib, filgotinib, lestaurtinib, pacritinib).
12. Participants who had an adequate response to JAK inhibitors will be excluded if the following are met:

    1. Use within 2 weeks prior to Baseline of topical JAK inhibitors.
    2. Use within 4 weeks prior to Baseline of systemic JAK inhibitors.
13. Use within 14 days prior to Baseline of: 1) systemic antibiotics, 2) calcipotriene or 3) retinoids.
14. Use within 7 days on the treatment area(s) prior to Baseline of: 1) topical antihistamines, 2) topical antibiotics, 3) topical corticosteroids or 4) other topical drug products.
15. Use of the following treatments prior to Baseline:

    1. For 5 half-lives or 12 weeks (whichever is longer) - biologic agents (e.g., dupilumab).
    2. For 4 weeks - systemic corticosteroids or adrenocorticotropic hormone analogs, cyclosporin, methotrexate, azathioprine, or other systemic immunosuppressive or immunomodulating agents (e.g., mycophenolate or tacrolimus).
    3. For 2 weeks - UVA/UVB therapy, PUVA (psoralen plus ultraviolet) therapy, tanning booths, or non-prescription UV light sources.
    4. For 2 weeks - immunizations and sedating antihistamines unless on long-term stable regimen (nonsedating antihistamines are permitted).
    5. For 2 weeks - use of other topical treatments for atopic dermatitis (other than bland emollients). Diluted sodium hypochlorite "bleach" baths are allowed if they do not exceed 2 baths per week and their frequency remains the same throughout the trial.
16. Uncontrolled systemic disease.
17. Any serious illness or condition(s) that, in the opinion of the PI, would interfere with full participation in the trial, including administration of IP and attending required trial visits; pose a significant risk to the participant; or interfere with interpretation of trial data.
18. Foreseen unprotected and intense/excessive UV exposure during the trial.
19. Scheduled or planned surgical procedures during the trial.
20. Unable or unwilling to comply with any of the trial requirements.
21. Medical or psychiatric conditions, or a personal situation, that may increase the risk associated with trial participation or may interfere with interpretation of trial results or participant compliance and, in the opinion of the PI, makes the participant inappropriate for trial entry.
22. Clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability.
23. Employees of the research center or Investigator.
24. Family of members of employees of the research center or Investigator.
25. Participants (e.g. siblings, spouses, relatives, roommates) residing in the same household cannot be enrolled at the same time.

    -

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | From enrollment to end of study at 8 weeks
  • Overall Incidence of safety events tabulated using the current version of the medical dictionary for regulatory activities (MedDRA).
evaluate effectiveness | From enrollment to end of study at 8 weeks
  Primary Efficacy Endpoint
  • Proportion of participants achieving Investigator's Global Assessment (IGA) response of "Clear" (Score 0) or "Almost Clear" (Score 1) with ≥ 2 grade of improvement at Week 8.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Center for Dermatology Clinical Research Inc., Fremont, California
  - Ablon Skin Institute and Research Center, Manhattan Beach, California
  - TCR Medical Corporation, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - USA and International Research Inc., Doral, Florida
  - FXM Clinical Research, Fort Lauderdale, Florida
  - Driven Research, Gables, Florida
  - FXM Clinical Research Miami, LLC, Miami, Florida
  - FXM Clinical Research Miramar, LLC, Miramar, Florida
  - Cordova Research Institute, Sweetwater, Florida
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - J&S Studies, Inc., New Brighton, Minnesota
  - JDR Dermatology Research, Las Vegas, Nevada
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch, Austin, Texas

IPD SHARING:
Plan to Share IPD: Undecided